CLINICAL TRIAL: NCT03249363
Title: Intraoperative Disinfection by Pulse Irrigation With Povidone-Iodine Solution in Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Gabriele Bernardi, MD, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: URome
Record Dates: First submitted 2017-07-05; First posted 2017-08-15 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Spinal Diseases; Spinal Fusion; Spine Injury; Infection, Hospital
Keywords: Pulse Irrigation Povidone Iodine Spine Surgery
MeSH Terms: conditions — Spinal Diseases; Spinal Injuries; Cross Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Pulsed PVP-I Irrigation (Experimental): Group in wich the patients who underwent spinal surgery were treated with 5-10 minutes of low-pressure irrigation with Povidone-Iodine (PVP-I) diluted to a 3% concentration (30g/l) in 2 l of saline performed before applying the bone graft
  Interventions: Procedure: Group A - Pulsed PVP-I Irrigation
- Group B - Pulsed Saline Irrigation (Active Comparator): Group in wich the patients who underwent spinal surgery were treated with 5-10 minutes of low-pressure irrigation with only 2 litres of saline solution (without povidone Iodine) performed before applying the bone graft
  Interventions: Procedure: Group A - Pulsed PVP-I Irrigation

INTERVENTIONS:
Procedure: Group A - Pulsed PVP-I Irrigation

SUMMARY:
The purpose of this study was to evaluate the efficacy, in preventing Spinal Surgical Infection, of intraoperative pulsatile irrigation with a 2000-ml saline solution of PVP-Iodine in a group of patients undergoing complex spine surgery with a posterior approach. To confirm and better assess the efficacy of intraoperative irrigation on the infection rate in spinal surgery, specimens for bacterial culture were harvested by swabs from muscular tissue before and after irrigation of the wounds

DETAILED DESCRIPTION:
The investigators enrolled fifty patients undergoing spinal surgery were randomly divided in two subgroups (A and B) of 25 patients each. In subgroup A, wounds were irrigated with dilute (3%) povidone-iodine solution through a low-pressure pulsatile device. In subgroup B wounds were irrigated with normal saline solution thorough a bulb syringe. In both subgroup specimens for bacterial culture were harvested by swabs from surgical site before and after irrigation of the wounds.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Patients candidated to spinal surgery for spinal surgery
* Primary spinal surgery procedure

Exclusion Criteria:

* Clinical signs of infection before surgery
* Previous spinal surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With surgical site infection | From the surgery to 1 year after
  Comparison of the results obtained from microbiological bacterial cultures of samples harvested during complex spine surgery in two groups of patients treated intraoperatively with pulsatile irrigation with diluted PVP-I (group A) or pulsatile irrigation with saline solution (group B)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schuster JM, Rechtine G, Norvell DC, Dettori JR. The influence of perioperative risk factors and therapeutic interventions on infection rates after spine surgery: a systematic review. Spine (Phila Pa 1976). 2010 Apr 20;35(9 Suppl):S125-37. doi: 10.1097/BRS.0b013e3181d8342c. PMID 20407344
- [Background] National Nosocomial Infections Surveillance (NNIS) System Report, Data Summary from January 1992-June 2001, issued August 2001. Am J Infect Control. 2001 Dec;29(6):404-21. doi: 10.1067/mic.2001.119952. No abstract available. PMID 11743489
- [Background] Watters WC 3rd, Baisden J, Bono CM, Heggeness MH, Resnick DK, Shaffer WO, Toton JF; North American Spine Society. Antibiotic prophylaxis in spine surgery: an evidence-based clinical guideline for the use of prophylactic antibiotics in spine surgery. Spine J. 2009 Feb;9(2):142-6. doi: 10.1016/j.spinee.2008.05.008. Epub 2008 Jul 10. PMID 18619911
- [Background] Barker FG 2nd. Efficacy of prophylactic antibiotic therapy in spinal surgery: a meta-analysis. Neurosurgery. 2002 Aug;51(2):391-400; discussion 400-1. PMID 12182777
- [Background] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists; Infectious Disease Society of America; Surgical Infection Society; Society for Healthcare Epidemiology of America. Clinical practice guidelines for antimicrobial prophylaxis in surgery. Am J Health Syst Pharm. 2013 Feb 1;70(3):195-283. doi: 10.2146/ajhp120568. No abstract available. PMID 23327981
- [Background] Sansur CA, Smith JS, Coe JD, Glassman SD, Berven SH, Polly DW Jr, Perra JH, Boachie-Adjei O, Shaffrey CI. Scoliosis research society morbidity and mortality of adult scoliosis surgery. Spine (Phila Pa 1976). 2011 Apr 20;36(9):E593-7. doi: 10.1097/BRS.0b013e3182059bfd. PMID 21325989
- [Background] Tsirikos AI, Lipton G, Chang WN, Dabney KW, Miller F. Surgical correction of scoliosis in pediatric patients with cerebral palsy using the unit rod instrumentation. Spine (Phila Pa 1976). 2008 May 1;33(10):1133-40. doi: 10.1097/BRS.0b013e31816f63cf. PMID 18449049
- [Background] Sponseller PD, LaPorte DM, Hungerford MW, Eck K, Bridwell KH, Lenke LG. Deep wound infections after neuromuscular scoliosis surgery: a multicenter study of risk factors and treatment outcomes. Spine (Phila Pa 1976). 2000 Oct 1;25(19):2461-6. doi: 10.1097/00007632-200010010-00007. PMID 11013497
- [Background] Epstein NE. Do silver-impregnated dressings limit infections after lumbar laminectomy with instrumented fusion? Surg Neurol. 2007 Nov;68(5):483-5; discussion 485. doi: 10.1016/j.surneu.2007.05.045. PMID 17961738
- [Background] Lu M, Hansen EN. Hydrogen Peroxide Wound Irrigation in Orthopaedic Surgery. J Bone Jt Infect. 2017 Jan 1;2(1):3-9. doi: 10.7150/jbji.16690. eCollection 2017. PMID 28529858
- [Background] Gruenberg MF, Campaner GL, Sola CA, Ortolan EG. Ultraclean air for prevention of postoperative infection after posterior spinal fusion with instrumentation: a comparison between surgeries performed with and without a vertical exponential filtered air-flow system. Spine (Phila Pa 1976). 2004 Oct 15;29(20):2330-4. doi: 10.1097/01.brs.0000142436.14735.53. PMID 15480149
- [Background] Celik SE, Kara A. Does shaving the incision site increase the infection rate after spinal surgery? Spine (Phila Pa 1976). 2007 Jul 1;32(15):1575-7. doi: 10.1097/BRS.0b013e318074c39f. PMID 17621202
- [Background] Rogers DM, Blouin GS, O'Leary JP. Povidone-iodine wound irrigation and wound sepsis. Surg Gynecol Obstet. 1983 Nov;157(5):426-30. PMID 6635913
- [Background] Brandt C, Hott U, Sohr D, Daschner F, Gastmeier P, Ruden H. Operating room ventilation with laminar airflow shows no protective effect on the surgical site infection rate in orthopedic and abdominal surgery. Ann Surg. 2008 Nov;248(5):695-700. doi: 10.1097/SLA.0b013e31818b757d. PMID 18948793
- [Background] Viljanto J. Disinfection of surgical wounds without inhibition of normal wound healing. Arch Surg. 1980 Mar;115(3):253-6. doi: 10.1001/archsurg.1980.01380030009003. PMID 7356379
- [Background] Lineaweaver W, McMorris S, Soucy D, Howard R. Cellular and bacterial toxicities of topical antimicrobials. Plast Reconstr Surg. 1985 Mar;75(3):394-6. doi: 10.1097/00006534-198503000-00016. PMID 3975287
- [Background] Crowley DJ, Kanakaris NK, Giannoudis PV. Irrigation of the wounds in open fractures. J Bone Joint Surg Br. 2007 May;89(5):580-5. doi: 10.1302/0301-620X.89B5.19286. PMID 17540739
- [Background] Anglen JO. Wound irrigation in musculoskeletal injury. J Am Acad Orthop Surg. 2001 Jul-Aug;9(4):219-26. doi: 10.5435/00124635-200107000-00001. PMID 11476531
- [Background] Jarvis WR, Edwards JR, Culver DH, Hughes JM, Horan T, Emori TG, Banerjee S, Tolson J, Henderson T, Gaynes RP, et al. Nosocomial infection rates in adult and pediatric intensive care units in the United States. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):185S-191S. doi: 10.1016/0002-9343(91)90367-7. PMID 1928163
- [Background] Culver DH, Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG, Banerjee SN, Edwards JR, Tolson JS, Henderson TS, et al. Surgical wound infection rates by wound class, operative procedure, and patient risk index. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):152S-157S. doi: 10.1016/0002-9343(91)90361-z. PMID 1656747
- [Background] McGirt MJ, Parker SL, Lerner J, Engelhart L, Knight T, Wang MY. Comparative analysis of perioperative surgical site infection after minimally invasive versus open posterior/transforaminal lumbar interbody fusion: analysis of hospital billing and discharge data from 5170 patients. J Neurosurg Spine. 2011 Jun;14(6):771-8. doi: 10.3171/2011.1.SPINE10571. Epub 2011 Mar 18. PMID 21417699
- [Background] Kaye KS, Anderson DJ, Sloane R, Chen LF, Choi Y, Link K, Sexton DJ, Schmader KE. The effect of surgical site infection on older operative patients. J Am Geriatr Soc. 2009 Jan;57(1):46-54. doi: 10.1111/j.1532-5415.2008.02053.x. PMID 19054183
- [Background] Weber WP, Zwahlen M, Reck S, Feder-Mengus C, Misteli H, Rosenthal R, Brandenberger D, Oertli D, Widmer AF, Marti WR. Economic burden of surgical site infections at a European university hospital. Infect Control Hosp Epidemiol. 2008 Jul;29(7):623-9. doi: 10.1086/589331. PMID 18564917
- [Background] Calderone RR, Garland DE, Capen DA, Oster H. Cost of medical care for postoperative spinal infections. Orthop Clin North Am. 1996 Jan;27(1):171-82. PMID 8539047
- [Background] Goldenheim PD. In vitro efficacy of povidone-iodine solution and cream against methicillin-resistant Staphylococcus aureus. Postgrad Med J. 1993;69 Suppl 3:S62-5. PMID 8290460
- [Background] Block C, Robenshtok E, Simhon A, Shapiro M. Evaluation of chlorhexidine and povidone iodine activity against methicillin-resistant Staphylococcus aureus and vancomycin-resistant Enterococcus faecalis using a surface test. J Hosp Infect. 2000 Oct;46(2):147-52. doi: 10.1053/jhin.2000.0805. PMID 11049709
- [Background] Perencevich EN, Sands KE, Cosgrove SE, Guadagnoli E, Meara E, Platt R. Health and economic impact of surgical site infections diagnosed after hospital discharge. Emerg Infect Dis. 2003 Feb;9(2):196-203. doi: 10.3201/eid0902.020232. PMID 12603990
- [Background] Hill RL, Casewell MW. The in-vitro activity of povidone-iodinecream against Staphylococcus aureus and its bioavailability in nasal secretions. J Hosp Infect. 2000 Jul;45(3):198-205. doi: 10.1053/jhin.2000.0733. PMID 10896798
- [Background] McLure AR, Gordon J. In-vitro evaluation of povidone-iodine and chlorhexidine against methicillin-resistant Staphylococcus aureus. J Hosp Infect. 1992 Aug;21(4):291-9. doi: 10.1016/0195-6701(92)90139-d. PMID 1355784
- [Background] van Meurs SJ, Gawlitta D, Heemstra KA, Poolman RW, Vogely HC, Kruyt MC. Selection of an optimal antiseptic solution for intraoperative irrigation: an in vitro study. J Bone Joint Surg Am. 2014 Feb 19;96(4):285-91. doi: 10.2106/JBJS.M.00313. PMID 24553884
- [Background] Kaysinger KK, Nicholson NC, Ramp WK, Kellam JF. Toxic effects of wound irrigation solutions on cultured tibiae and osteoblasts. J Orthop Trauma. 1995;9(4):303-11. doi: 10.1097/00005131-199509040-00006. PMID 7562152
- [Background] Bhandari M, Schemitsch EH, Adili A, Lachowski RJ, Shaughnessy SG. High and low pressure pulsatile lavage of contaminated tibial fractures: an in vitro study of bacterial adherence and bone damage. J Orthop Trauma. 1999 Nov;13(8):526-33. doi: 10.1097/00005131-199911000-00002. PMID 10714777
- [Background] Dirschl DR, Duff GP, Dahners LE, Edin M, Rahn BA, Miclau T. High pressure pulsatile lavage irrigation of intraarticular fractures: effects on fracture healing. J Orthop Trauma. 1998 Sep-Oct;12(7):460-3. doi: 10.1097/00005131-199809000-00005. PMID 9781768
- [Background] Flow Investigators. Fluid lavage of open wounds (FLOW): design and rationale for a large, multicenter collaborative 2 x 3 factorial trial of irrigating pressures and solutions in patients with open fractures. BMC Musculoskelet Disord. 2010 May 6;11:85. doi: 10.1186/1471-2474-11-85. PMID 20459600
- [Background] Abdul-Jabbar A, Berven SH, Hu SS, Chou D, Mummaneni PV, Takemoto S, Ames C, Deviren V, Tay B, Weinstein P, Burch S, Liu C. Surgical site infections in spine surgery: identification of microbiologic and surgical characteristics in 239 cases. Spine (Phila Pa 1976). 2013 Oct 15;38(22):E1425-31. doi: 10.1097/BRS.0b013e3182a42a68. PMID 23873240
- [Derived] De Luna V, Mancini F, De Maio F, Bernardi G, Ippolito E, Caterini R. Intraoperative Disinfection by Pulse Irrigation with Povidone-Iodine Solution in Spine Surgery. Adv Orthop. 2017;2017:7218918. doi: 10.1155/2017/7218918. Epub 2017 Oct 2. PMID 29098088